CLINICAL TRIAL: NCT00229528
Title: Dose Ranging Study of the Effect of Paroxetine on COAT-Platelet Production in Normal Volunteers and Patients With Cardiovascular Disease
Brief Title: Effect of Paroxetine on COAT-Platelet Production in Normal Volunteers and Patients With Cardiovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Stephen Hamilton, University of Oklahoma Dept of Pharmacy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000774
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Paroxetine

INTERVENTIONS:
Drug: Paxil-CR

SUMMARY:
COAT-platelets stands for collagen and thrombin stimulated platelets, which are two things in the body that make platelets stick together. These platelets may be important in the initiation of a heart attack (myocardial infarction). A chemical in the body called serotonin maybe responsible for COAT-platelet production. Paroxetine causes a significant reduction in platelet serotonin and therefore may have value in preventing heart attacks. Therefore, the current study is designed to determine whether paroxetine will decrease COAT-platelet production in normal volunteers and patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* normal volunteers (without heart disease)
* patients with heart disease
* between ages 18 & 65

Exclusion Criteria:

* children less than 18 years
* adults greater than 65 years
* those who can not keep appointments
* patients within 2 weeks of a coronary catheterization
* patients within 6 months of unstable angina or myocardial infarction
* individuals with allergies to paroxetine or similar medications
* individuals having adverse events to paroxetine or similar medications
* individuals with diagnosis of mania
* individuals with a diagnosis of hypomania
* individuals with a diagnosis of bipolar disorders
* individuals with a diagnosis of depression
* individuals with a diagnosis of panic disorders
* individuals with a diagnosis of seizure disorders
* individuals with a history of suicide attempts
* individuals with a diagnosis of hyponatremia
* individuals with active bleeding disorders
* individuals with a diagnosis of narrow angle glaucoma
* individuals with an estimated creatinine clearance of less that 30 ml/min
* individuals taking potentially interacting medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To define the percent COAT-platelet and response to Paxil-CR in 5 control subjects.

SECONDARY OUTCOMES:
To define the percent COAT-platelet and response to Paxil-CR in 20 patients with Coronary Artery Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F. Hamilton, Pharm.D., Principal Investigator — The University of Oklahoma College of Pharmacy
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States